CLINICAL TRIAL: NCT01868724
Title: Identification and Validation of Biomarkers of Acute Kidney Injury Recovery
Status: Completed | Type: Observational
Sponsor: Astute Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Ruby
Record Dates: First submitted 2013-05-21; First posted 2013-06-04 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2014-09

CONDITIONS: Acute Kidney Injury
Keywords: Kidney Renal
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is to collect blood and urine samples to help identify and validate protein biomarkers of recovery from moderate or severe acute kidney injury (AKI).

ELIGIBILITY:
Inclusion Criteria:a.

* Males and females 21 years of age or older
* Receiving care in an intensive care unit
* Expected to remain in the ICU for at least 48 hours after enrollment
* Use of indwelling urinary catheter as standard care at the time of enrollment
* Subject must have acute kidney injury (KDIGO stage 2 or stage 3) at the time of the first sample collection
* First sample must be collected within 36 hours of meeting KDIGO stage 2 criteria
* Written informed consent provided by patient or legally authorized representative (LAR)

Exclusion Criteria:

* Prior kidney transplantation
* Comfort-measures-only status
* Already receiving dialysis (either acute or chronic) or in imminent need of dialysis at the time of enrollment
* History of human immunodeficiency virus (HIV) or hepatitis virus (based upon available medical records) infections (NOTE: HIV or hepatitis testing need not be performed for enrollment in this study.)
* Special populations, pregnant women, prisoners or institutionalized individuals
* Patient meets any of the following:

  * Active bleeding with an anticipated need for > 4 units PRBC in a day
  * Hemoglobin < 7 g/dL
  * Any other condition that in the physician's opinion would contraindicate drawing serial blood samples for clinical study purposes

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult ICU Patients with AKI
Sampling Method: Non-Probability Sample
Enrollment: 362 (Actual)
Dates: Start 2013-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Validation of biomarkers for Acute Kidney Injury Recovery in Blood or Urine. | Day 1-7 of enrollment
  This study is a multi-center study intended to enroll enough subjects to validate biomarkers for acute kidney injury recovery. Subjects enrolled will be those with known moderate to severe AKI. The study is to determine the outcome of Major Adverse Kidney Event (MAKE) and Major Adverse Cardiac Event (MACE) during a period of up to 7 days.

SECONDARY OUTCOMES:
None at this time | 10 months
  There are no secondary outcomes measures planned at this time

CONTACTS AND LOCATIONS:
Overall Officials: Lakhmir S Chawla, M.D., Principal Investigator — George Washington University
Locations (18):
- United States (10):
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Chicago, Illinois
  - Baltimore, Massachusetts
  - Ann Arbor, Michigan
  - Durham, North Carolina
  - Akron, Ohio
  - Cleveland, Ohio
  - Pittsburgh, Pennsylvania
  - Nashville, Tennessee
- Innsbruck, Austria
- Belgium (2):
  - Brussels
  - Ghent
- Germany (2):
  - Frankfurt
  - Madgeburg
- Sabadelle, Spain
- United Kingdom (2):
  - London
  - West Sussex

REFERENCES:
- [Derived] Koyner JL, Chawla LS, Bihorac A, Gunnerson KJ, Schroeder R, Demirjian S, Hodgson L, Frey JA, Wilber ST, Kampf JP, Kwan T, McPherson P, Kellum JA; RUBY investigators. Performance of a Standardized Clinical Assay for Urinary C-C Motif Chemokine Ligand 14 (CCL14) for Persistent Severe Acute Kidney Injury. Kidney360. 2022 Mar 24;3(7):1158-1168. doi: 10.34067/KID.0008002021. eCollection 2022 Jul 28. PMID 35919538
- [Derived] Hoste E, Bihorac A, Al-Khafaji A, Ortega LM, Ostermann M, Haase M, Zacharowski K, Wunderink R, Heung M, Lissauer M, Self WH, Koyner JL, Honore PM, Prowle JR, Joannidis M, Forni LG, Kampf JP, McPherson P, Kellum JA, Chawla LS; RUBY Investigators. Identification and validation of biomarkers of persistent acute kidney injury: the RUBY study. Intensive Care Med. 2020 May;46(5):943-953. doi: 10.1007/s00134-019-05919-0. Epub 2020 Feb 6. PMID 32025755